CLINICAL TRIAL: NCT02212119
Title: A Randomized, Placebo Controlled Trial of Botulinum Toxin for Paratonic Rigidity in People With Advanced Cognitive Impairment
Brief Title: Safety and Effectiveness of Botulinum Toxin in Elderly Patients With Dementia and Muscle Stiffness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistive Technology Clinic, Canada (Other)
Collaborators: Merz Pharmaceuticals GmbH (Industry); Baycrest (Other)
Responsible Party: Principal Investigator, Dr. Galit Kleiner-Fisman, Medical Director, Assistive Technology Clinic, Assistant Professor Department of Medicine, University of Toronto, Assistive Technology Clinic, Canada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NT-036
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Dementia; Paratonia
Keywords: Dementia; Paratonia; Caregiver Burden; Botulinum toxin
MeSH Terms: conditions — Dementia; Muscle Rigidity; Caregiver Burden | interventions — Botulinum Toxins; incobotulinumtoxinA; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): Saline injection up to 5 cc in arm with paratonia (one time injection)
  Interventions: Drug: Saline
- Botulinum Toxin (Active Comparator): Up to 300 U (5 cc) of Botulinum toxin diluted 2:1 (2 cc per 100 U of Botulinum toxin) (one time injection)
  Interventions: Drug: Botulinum Toxin

INTERVENTIONS:
Drug: Botulinum Toxin
  Other Names: Xeomin
  Arms: Botulinum Toxin
Drug: Saline
  Arms: Saline

SUMMARY:
Aim of the study is to perform a pilot study to assess the impact of Botulinum toxin on muscle tone, and caregiver burden in individuals who are cognitively impaired and who are fully dependent.

The primary objective is to confirm proof of principle that paratonic rigidity and the consequences associated with it can be reduced with injection of Botulinum toxin injections resulting in reduced care-giver burden.

The secondary objectives are to determine optimal time points for evaluation of efficacy in this patient population and whether the time period is sufficient for washout of Botulinum toxin effect; determine most salient and sensitive outcome measures; identify obstacles in data gathering; and lastly, to determine feasibility of battery of assessments in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Severe cognitive impairment (complete dependency in all activities of daily living (ADLs)
* Diagnosis of Alzheimer's disease, vascular dementia,or frontotemporal dementia
* Score> 3 on the paratonic assessment instrument, with paratonic rigidity in an arm(s) interfering in the provision of care

Exclusion Criteria:

* Alternate etiologies for increased tone
* Botulinum toxin 6 months preceding the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2013-02 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Impact on care-giver burden | 6 weeks for primary outcome, 32 weeks for entire study
  Impact on caregiver burden in providing upper extremity care.
  Measured by the Carer Burden Scale which includes four items (cleaning the palm, cutting the fingernails, dressing, cleaning under the armpit).
  Each item rated on five point Likert scale ("no difficulty" to "cannot do task").

SECONDARY OUTCOMES:
Visual Analogue Scale | 6 weeks for secondary outcome, 32 weeks for entire study
  Completed by the professional caregiver that is caring for the patient to assess perception of ease of caregiving.
  Consists of 100 mm line with anchors of 0 "giving care to the residents is very difficult" and 100 "giving care to the residents is very easy"
Joint angle measurement | 6 weeks for secondary outcome, 32 weeks for entire study
  Joint angle measurements were used reflecting range of motion.
  Used as a surrogate measure for severity of paratonia
Pain | 6 weeks for secondary outcome, 32 weeks for entire study
  Pain Assessment in Advanced Dementia (PAINAD) Scale used to evaluate correlates of pain and determine whether Botulinum toxin treatment reduces discomfort of morning care.
  Consists of 5 items (breathing, negative vocalization, facial expression, body language and consolability), scored on a 0-2 point scale and then summed to arrive at a total scale.
Global Assessment | 6 weeks for secondary outcome, 32 weeks for entire study
  Overall response to treatment evaluated by study investigator and by professional caregiver caring for patient using the global assessment scale.
  A score of -4 indicates very marked worsening, 0 no change, and +4 very marked improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Galit Kleiner-Fisman, MD, Principal Investigator — University of Toronto, Baycrest
Locations (1):
- Assistive Technology Clinic at Baycrest, Toronto, Ontario, Canada

REFERENCES:
- [Background] Canadian study of health and aging: study methods and prevalence of dementia. CMAJ. 1994 Mar 15;150(6):899-913. PMID 8131123
- [Background] Matthews FE, Dening T; UK Medical Research Council Cognitive Function and Ageing Study. Prevalence of dementia in institutional care. Lancet. 2002 Jul 20;360(9328):225-6. doi: 10.1016/S0140-6736(02)09461-8. PMID 12133659
- [Background] Fox PJ, Kohatsu N, Max W, Arnsberger P. Estimating the costs of caring for people with Alzheimer disease in California: 2000-2040. J Public Health Policy. 2001;22(1):88-97. PMID 11382092
- [Background] Hobbelen JS, Koopmans RT, Verhey FR, Habraken KM, de Bie RA. Diagnosing paratonia in the demented elderly: reliability and validity of the Paratonia Assessment Instrument (PAI). Int Psychogeriatr. 2008 Aug;20(4):840-52. doi: 10.1017/S1041610207006424. Epub 2008 Jan 7. PMID 18177542
- [Background] Franssen EH, Kluger A, Torossian CL, Reisberg B. The neurologic syndrome of severe Alzheimer's disease. Relationship to functional decline. Arch Neurol. 1993 Oct;50(10):1029-39. doi: 10.1001/archneur.1993.00540100024010. PMID 8215960
- [Background] Hobbelen JS, Verhey FR, Bor JH, de Bie RA, Koopmans RT. Passive movement therapy in patients with moderate to severe paratonia; study protocol of a randomised clinical trial (ISRCTN43069940). BMC Geriatr. 2007 Dec 19;7:30. doi: 10.1186/1471-2318-7-30. PMID 18093298
- [Background] Souren LE, Franssen EH, Reisberg B. Neuromotor changes in Alzheimer's disease: implications for patient care. J Geriatr Psychiatry Neurol. 1997 Jul;10(3):93-8. doi: 10.1177/089198879701000301. PMID 9322130
- [Background] Kao I, Drachman DB, Price DL. Botulinum toxin: mechanism of presynaptic blockade. Science. 1976 Sep 24;193(4259):1256-8. doi: 10.1126/science.785600.
- [Background] Brashear A, Gordon MF, Elovic E, Kassicieh VD, Marciniak C, Do M, Lee CH, Jenkins S, Turkel C; Botox Post-Stroke Spasticity Study Group. Intramuscular injection of botulinum toxin for the treatment of wrist and finger spasticity after a stroke. N Engl J Med. 2002 Aug 8;347(6):395-400. doi: 10.1056/NEJMoa011892. PMID 12167681
- [Background] Elovic EP, Brashear A, Kaelin D, Liu J, Millis SR, Barron R, Turkel C. Repeated treatments with botulinum toxin type a produce sustained decreases in the limitations associated with focal upper-limb poststroke spasticity for caregivers and patients. Arch Phys Med Rehabil. 2008 May;89(5):799-806. doi: 10.1016/j.apmr.2008.01.007. PMID 18452724
- [Background] Giovannelli M, Borriello G, Castri P, Prosperini L, Pozzilli C. Early physiotherapy after injection of botulinum toxin increases the beneficial effects on spasticity in patients with multiple sclerosis. Clin Rehabil. 2007 Apr;21(4):331-7. doi: 10.1177/0269215507072772. PMID 17613573
- [Background] Simpson DM, Gracies JM, Yablon SA, Barbano R, Brashear A; BoNT/TZD Study Team. Botulinum neurotoxin versus tizanidine in upper limb spasticity: a placebo-controlled study. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):380-5. doi: 10.1136/jnnp.2008.159657. Epub 2008 Oct 31. PMID 18977811
- [Background] Wells DL, Dawson P, Sidani S, Craig D, Pringle D. Effects of an abilities-focused program of morning care on residents who have dementia and on caregivers. J Am Geriatr Soc. 2000 Apr;48(4):442-9. doi: 10.1111/j.1532-5415.2000.tb04704.x. PMID 10798473
- [Background] Brin MF. Dosing, administration, and a treatment algorithm for use of botulinum toxin A for adult-onset spasticity. Spasticity Study Group. Muscle Nerve Suppl. 1997;6:S208-20. doi: 10.1002/(sici)1097-4598(1997)6+3.0.co;2-1. PMID 9826992
- [Background] Bhakta BB, Cozens JA, Chamberlain MA, Bamford JM. Impact of botulinum toxin type A on disability and carer burden due to arm spasticity after stroke: a randomised double blind placebo controlled trial. J Neurol Neurosurg Psychiatry. 2000 Aug;69(2):217-21. doi: 10.1136/jnnp.69.2.217. PMID 10896696
- [Background] Warden V, Hurley AC, Volicer L. Development and psychometric evaluation of the Pain Assessment in Advanced Dementia (PAINAD) scale. J Am Med Dir Assoc. 2003 Jan-Feb;4(1):9-15. doi: 10.1097/01.JAM.0000043422.31640.F7. PMID 12807591
- [Background] Naumann M, Yakovleff A, Durif F; BOTOX Cervical Dystonia Prospective Study Group. A randomized, double-masked, crossover comparison of the efficacy and safety of botulinum toxin type A produced from the original bulk toxin source and current bulk toxin source for the treatment of cervical dystonia. J Neurol. 2002 Jan;249(1):57-63. doi: 10.1007/pl00007848. PMID 11954869
- [Background] Albright AL, Barron WB, Fasick MP, Polinko P, Janosky J. Continuous intrathecal baclofen infusion for spasticity of cerebral origin. JAMA. 1993 Nov 24;270(20):2475-7. PMID 8230625
- [Background] Smetanin P, Kobak P, Briante C, Ahmad S. Rising Tide: The Impact of Dementia in Canada 2008 to 2038. RiskAnalytica; 2009.
- [Background] Knapp M, Comas-Herrera, Somani A, Banerjee S. Dementia: Summary report for the National Audit Office international comparisons. London: Personal Social Services Research Unit London School of Economics and Political Science and Section of Mental Health and Ageing The Institute of Psychiatry, King's College London; 2007.
- [Background] Dupre E. Debilite mentale and debilite motrice associees. Rev Neurol 1910;20:54-56.
- [Background] Delagi EF, Perotto A, Iazzetti J, Morrison D. Anatomic Guides for the Elecromyographer. In: Charles C.Thomas, ed., 2nd ed Springfield, 1980.
- [Background] Bhakta BB, Tennant A, Cozens JA, et al. Application of item response theory to measure the disabling effects of severe upper limb spasticity in stroke and the consequent carer burden. Cerebrovascular Dis 1999;9:124.
- [Background] Waltz CFSOL, Lenz ER. Measurement in Nursing Research, 2nd ed. Philadelphia: F.A. Davis, 1991.
- [Background] Waardenburg H, Elvers W, Van Vechgel F, Oostendorp R. Can paratonia be measured reliably? Evaluation of the reliability of a visual analogue scale and the modified tonus sclae of Ashworth for measuring paratonia. Nederlands Tijdschrift voor Fysiotherapie (in dutch) 1999;102:30-35.
- [Derived] Kleiner-Fisman G, Khoo E, Moncrieffe N, Forbell T, Gryfe P, Fisman D. A randomized, placebo controlled pilot trial of botulinum toxin for paratonic rigidity in people with advanced cognitive impairment. PLoS One. 2014 Dec 23;9(12):e114733. doi: 10.1371/journal.pone.0114733. eCollection 2014. PMID 25536218